CLINICAL TRIAL: NCT05009498
Title: Vitamin D3 Supplementation vs Placebo for Vitamin D Deficient/Insufficient Patients Undergoing Arthroscopic Rotator Cuff Repair: a Quadruple-blinded Randomized Controlled Trial
Brief Title: Vitamin D3 Supplementation for Vitamin D Deficiency in Rotator Cuff Repair Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Community Memorial Health System (Other)
Responsible Party: Principal Investigator, Michael Bogard, Orthopedic Surgery Resident, Community Memorial Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VITD3RCR
Record Dates: First submitted 2021-07-23; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Vitamin D Deficiency; Rotator Cuff Tears
Keywords: Rotator Cuff repair; Rotator Cuff tears; Vitamin D deficiency; Vitamin D3 supplementation; Shoulder arthroscopy
MeSH Terms: conditions — Vitamin D Deficiency; Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization at the level of the manufacturer, therefore all patients, investigators, care providers and outcomes assessors with be blinded throughout the duration of the investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Patient will receive a placebo dosing, identical in appearance and at the same intervals as the interventional dose
  Interventions: Other: Placebo
- Vitamin D3 supplementation group (Active Comparator): Patient will receive high-dose Vitamin D3 supplementation in capsule form, identical in appearance and at the same intervals as the placebo dose
  Interventions: Dietary Supplement: Vitamin D3 supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin D3 supplementation — Vitamin D3 in 50,000 IU capsules Loading dose of 150,000 IUs (3 capsules) Interval dosing of 50,000 IUs (1 capsule) every 2 weeks for 1 year
  Arms: Vitamin D3 supplementation group
Other: Placebo — Placebo capsule, identical in appearance to the Vitamin D3 supplement capsule Dosing intervals identical in duration and quantity as Vitamin D3 supplement group
  Arms: Placebo group

SUMMARY:
Rotator cuff injuries are the most common cause of shoulder disability and is increasingly more prevalent in the aging population. Rotator cuff repair has long been the mainstay of treatment for symptomatic full-thickness tears and medium to large partial thickness tears that do no improve with nonoperative therapies.

Approximately 32% of the US population is Vitamin D deficient. This is important for many health reasons, but specifically, Vitamin D has been found to play a critical role in bone mineralization and fracture healing/prevention. There is emerging data to support Vitamin D's role in regulating the inflammatory response throughout the body, which includes soft tissue (i.e. tendons) healing. The role of Vitamin D in tendon to bone healing has yet to be fully investigated, yet it is reasonable to conclude that normal blood levels of Vitamin D would optimize the setting for healing in rotator cuff repair.

The investigators hypothesize that Vitamin D deficient patients undergoing shoulder rotator cuff repair will experience more positive outcomes and decreased complications when supplemented with Vitamin D3, compared to Vitamin D deficient patients who do not receive supplementation. The objective of this study is to demonstrate the positive effect of Vitamin D3 in rotator cuff repair healing and patient reported outcomes in patients who are Vitamin D deficient

DETAILED DESCRIPTION:
Rotator cuff pathology is the most common cause of shoulder disability and is increasingly more prevalent in the aging population. Incidence increases in a direct relationship to age. It is reported that over the age of 60, 28% of patients had full-thickness tears and 26% had partial thickness tears. Increasing age, history of trauma and hand dominance are associated risk factors for rotator cuff tearing. Rotator cuff tears (RCT) can occur from a degenerative process that increases with age, but also associated with micro- or macrotrauma. Rotator cuff repair (RCR) has long been the mainstay treatment for symptomatic full-thickness tears and medium to large partial thickness tears that have failed conservative measures. Long term clinical results for rotator cuff repair exceed 90% good to excellent results at 10 years.

According to the National Center for Health Statistics, approximately 32% of the US population is Vitamin D deficient. It has been widely accepted and studied that Vitamin D (25OHD) plays an important role in bone mineralization and fracture healing/prevention. Also, numerous studies have discovered the association of Vitamin D insufficiency with non-skeletal conditions such as Type 2 diabetes mellitus, cardiovascular disease, chronic pulmonary disease, tuberculosis, and upper respiratory conditions. There is an emerging focus on the role of Vitamin D and soft tissue healing and function.

Vitamin D decreases inflammation in the body by downregulating TNF alpha, which in turn decreases the amount of MMP-9 secreted. Increased MMPs have been associated with poor healing in rotator cuff muscles. Vitamin D levels have also been shown to affect the expression of BMPs, TGF-beta, and RANK.

Vitamin D receptors have been discovered on important soft tissue structures including tendons. It has been posited that Vitamin D's effect on regulating the inflammatory response is associated with tendon healing and overall function.

Traditional oral dosing for Vitamin D is in the Vitamin D3 form. Dosing quantities range from 400 IU to 5000 IU/day. In significantly deficient patients, it is not uncommon to see 50,000 IU/week for several weeks to achieve normal serum Vitamin D levels.

Studies have shown that the human body will generate up to 10,000-25,000 IU/day from sun exposure. This finding, among others, has called into question the arbitrary values set by IOM/ES to quantify serum levels for Vitamin D sufficient, insufficiency, or deficiency. Also, the daily recommended dosing quantities.

Vitamin D repletion therapy has been shown to be effective but often over protracted courses with no distinct linear relationship with the current recommendations set by the IOM/ES. Kerns et al 2014 performed the most comprehensive meta-analysis review of single, high-dose vitamin D supplementation and subsequent efficacy and safety. Their conclusion was that single vitamin D dosing of > 200,000 IU was able to sustain mean 25(OH)D concentrations > 30 ng/mL and there were no adverse effects noted at doses < 200,000. They also showed in all studies that peak serum 25(OH)D occurred at days 3-7. Some studies that examined single dose of 100,000 IU failed to achieve a serum 25(OH)D level of sufficiency for patients with baseline 25(OH)D of < 20ng/mL, and there were some reported adverse effects in single dose quantities of 300,000 to 600,000 IU (possible increased fracture risk, elevated bone turnover, transient serum hypercalcemia (> 500,000), and GI irritability).

With the prevalence of RCT and Vitamin D deficiency in the population, it is only reasonable to conclude that addressing the underlying biochemical processes to enhance soft tissue healing would provide a more favorable environment in the setting of rotator cuff repair. Orthopedic surgeons seek to optimize patient care by exhausting all available, and albeit reasonable, controllable variables The investigators hypothesize that Vitamin D deficient patients undergoing shoulder rotator cuff repair will experience more positive outcomes and decreased complications when supplemented with Vitamin D3, compared to Vitamin D deficient patients who do not receive supplementation.

The objective of this study is to demonstrate the positive effect of Vitamin D3 supplementation in rotator cuff repair healing and patient reported outcomes in patients who are Vitamin D deficient.

This is a prospective, quadruple-blinded, randomized, placebo-controlled study to evaluate the feasibility and effect of Vitamin D3 supplementation in Vitamin D deficient patients undergoing rotator cuff repair. Patients will be randomized to one of two arms, either Vitamin D3 supplementation or placebo. Each patient will be given a loading dose of 150,000 IUs prior to surgery, and then a bi-monthly maintenance dose of 50,000 IUs for one year. The patients will be followed for a total of 24 months following surgery. Clinical evidence of rotator cuff repair and patient reported outcome measures will be evaluated by chart review and patient questionnaires. All post-operative standard of care practices including laboratory tests, imaging, and rehabilitation will also be collected.

Enrollment will close once enough patients have been enrolled to achieve a 95% power. The investigators expect the study to take 2-3 years to complete.

Patients that meet all of the inclusion criteria and none of the exclusion criteria will be approached by the investigators, informed of the study, and provided with an informed consent form (ICF). Ample time will be given to the patient to review the ICF form in it's entirely and ask the investigator any questions they may have. If the patient agrees to participate, the will be asked to sign the ICF and the investigator obtaining consent will countersign. Patients will receive a copy of the signed consent form for their records, and the ICF will be scanned into the patient's medical record. The original paper copy of the ICF will be stored in a locked cabinet in the investigator's office. No data will be collected prior to completion of the informed consent form.

Once consent has been obtained, each participant will be assigned a subject ID number (ex. Subject # XXX). Baseline data will then be collected from the patient and their medical chart. These data points include: demographics, medical history, injury details, and rotator cuff tear pattern and location. A baseline patient reported outcomes questionnaire will also be obtained.

Feasibility of this study will be assessed over 24 months. Vitamin D3 and placebo will be administered over the course of the first 12 months of the study. Supplementation will begin between 3 and 7 days prior to the day of surgery, depending on the pre-operative scheduled appointment and relation to the day of surgery. The study participants will be expected to store and administer their scheduled dosing as instructed by the study team. Reminders prompting the patient's scheduled dosing will be sent via text and/or email, depending on patient preference as indicated on the initial questionnaire.

The loading dose and first maintenance dose following surgery will be administered to the patient at the study site. The bottle will then be provided to the participant for their personal storage and they will be instructed to take one 50,000 IU capsule (or identical placebo) once every two weeks for a total of 25 weeks (one year of total supplementation).

To ensure compliance, the participant will be asked to bring their bottle with them to each follow-up visit. At the 12 month follow-up visit, the participants will return their bottle to either the investigator or clinical research coordinator. If the participant does not return the bottle, the clinical research coordinator will provide them with an envelope to return it via mail.

Pre-operative labs will be ordered as standard of care and the results will be collected from the medical chart. Laboratory tests to be drawn are a comprehensive metabolic panel (CMP), serum 25(OH)D level, and complete blood count (CBC).

The study protocol does not dictate the surgical technique. Based on the study's eligibility criteria, all participants must receive tear pattern specific arthroscopic rotator cuff repair utilizing the double row versus single row technique. The orientation and final repair construct will be determined intraoperatively to the discretion of the treating surgeon. Surgical debridement, biceps tenotomy with or without tenodesis, and other surgical procedures will be performed as indicated for the benefit of the patient.

Details of the surgical management of the patient's rotator cuff tear will be collected from the medical record. Post-operative laboratory tests will be drawn per standard of care and collected from the medical record.

Post-operative rehabilitation will consist of sling utilization starting from post-operative day zero through week six, as per standard of care. Patients will be instructed on early passive range of motion (ROM) exercises (i.e. pendulum exercises) that will begin at the discretion of the treating surgeon. A recent study from AJSM (Keener et al, 2014) demonstrated no significant difference between early passive ROM vs 6 weeks of sling immobilization. The patient will be instructed to avoid active ROM (aROM) of the operative shoulder for the first 6 weeks, but will be allowed to remove the sling for elbow/wrist/hand ROM and hygiene. Starting at week one, patients will begin formal outpatient physical therapy (PT) twice a week. From weeks 6-12 patients will begin PT guided initiated assisted active ROM and aROM of the shoulder. From months 3-4, initiated cuff, deltoid, and scapular stabilizer strengthening. From month 4 and on, patients will begin full activities between months 4 through 6 on the basis of individual progress.

Details of the patient's rehabilitation course will be collected from the medical record The investigator who is the operative orthopedic surgeon will monitor patient safety for each of their patients involved in the study. The surgeon will be responsible for reviewing adverse events, enrollment numbers, and medical compliance. All serious adverse events will be recorded and promptly submitted according to the appropriate hospital policy. All serious adverse events will also be promptly reported to the IRB as well.

Following completion of this study, participants may be un-blinded from their treatment group upon request.

The patient questionnaires will be the primary data collection tool for the study. Other data points will be collected from the electronic medical record. Data will be stored on an encrypted database on password protected computers at the study site, only accessible to the investigators and study personnel. Data will be recorded at the time of collection. Hardcopy questionnaires and informed consent forms will be retained for double verification in a locked cabinet only accessible to the study team.

Study documents will be held in strict confidence by the investigators and other study personnel, and all efforts will be made to maintain patient confidentiality as per standard HIPAA requirements. All data will be de-identified prior to dissemination.

In accordance with 42 CFR 164.530(j)(2), all study records will be securely retained by the investigators for a minimum of 6 years following completion of the study

ELIGIBILITY:
Inclusion Criteria:

* Acute or chronic rotator cuff tear
* Small to medium sized rotator cuff tear
* Rotator cuff tear which can be treated with arthroscopic RCR (single or double row technique)
* Serum 25(OH)D levels < 30 ng/mL

Exclusion Criteria:

* Massive rotator cuff tear that is inoperable or requires superior capsular reconstruction (SCR)
* Revision RCR
* Serum 25(OH)D levels ≥ 30 ng/mL
* Elevated serum calcium (> 10.5 mg/dL)
* Known or likely undiagnosed disorders of bone metabolism (i.e. Pagets, ostemalacia, osteopetrosis, OI, etc.)
* History of hyperhomocysteinemia
* Vitamin D allergy or other contraindication to Vitamin D supplementation
* Patients currently taking OTC multivitamin that contains Vitamin and unwilling/unable to discontinue use for the duration of this study
* Patient who are pregnant or plan to become pregnant in the next two years
* In the judgment of the investigators, patients who will have trouble adhering to the study follow-up schedule or dosing schedule

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
University of California-Los Angeles Shoulder score | Baseline (Preop)
  Shoulder scoring system mainly consisting of two parts. Patients subjectively evaluate pain and functional activity; and doctors objectively evaluate shoulder joint range of motion and muscle strength. Scores range from 0 to 35, with a higher score indicating a better function.
Constant-Murray Shoulder Score | Baseline (Preop)
  Shoulder score system mainly consisting of two parts. Patients subjectively evaluate pain and activity level; doctors objectively evaluate shoulder joint range of motion and muscle strength. Scores range from 0 to 100, higher score indicating better function. Compare to contralateral (unaffected shoulder).
American Shoulder and Elbow Surgeon score | Baseline (Preop)
  Evaluation criteria used to assess shoulder joint function based on the patient's pain and accumulated daily activities. Possible scores range from 0 to 100, higher scores indicating better shoulder function.
SF-12 (12-item Short Form Survey) | Baseline (Preop)
  A general health questionnaire, drawn from the original SF-36 questionnaire. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average
University of California-Los Angeles Shoulder score | 6 weeks post op
  Shoulder scoring system mainly consisting of two parts. Patients subjectively evaluate pain and functional activity; and doctors objectively evaluate shoulder joint range of motion and muscle strength. Scores range from 0 to 35, with a higher score indicating a better function.
Constant-Murray Shoulder Score | 6 weeks post op
  Shoulder score system mainly consisting of two parts. Patients subjectively evaluate pain and activity level; doctors objectively evaluate shoulder joint range of motion and muscle strength. Scores range from 0 to 100, higher score indicating better function. Compare to contralateral (unaffected shoulder).
American Shoulder and Elbow Surgeon score | 6 weeks post op
  Evaluation criteria used to assess shoulder joint function based on the patient's pain and accumulated daily activities. Possible scores range from 0 to 100, higher scores indicating better shoulder function.
SF-12 (12-item Short Form Survey) | 6 weeks post op
  A general health questionnaire, drawn from the original SF-36 questionnaire. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average
University of California-Los Angeles Shoulder score | 12 weeks post op
  Shoulder scoring system mainly consisting of two parts. Patients subjectively evaluate pain and functional activity; and doctors objectively evaluate shoulder joint range of motion and muscle strength. Scores range from 0 to 35, with a higher score indicating a better function.
Constant-Murray Shoulder Score | 12 weeks post op
  Shoulder score system mainly consisting of two parts. Patients subjectively evaluate pain and activity level; doctors objectively evaluate shoulder joint range of motion and muscle strength. Scores range from 0 to 100, higher score indicating better function. Compare to contralateral (unaffected shoulder).
American Shoulder and Elbow Surgeon score | 12 weeks post op
  Evaluation criteria used to assess shoulder joint function based on the patient's pain and accumulated daily activities. Possible scores range from 0 to 100, higher scores indicating better shoulder function.
SF-12 (12-item Short Form Survey) | 12 weeks post op
  A general health questionnaire, drawn from the original SF-36 questionnaire. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average
University of California-Los Angeles Shoulder score | 6 months post op
  Shoulder scoring system mainly consisting of two parts. Patients subjectively evaluate pain and functional activity; and doctors objectively evaluate shoulder joint range of motion and muscle strength. Scores range from 0 to 35, with a higher score indicating a better function.
Constant-Murray Shoulder Score | 6 months post op
  Shoulder score system mainly consisting of two parts. Patients subjectively evaluate pain and activity level; doctors objectively evaluate shoulder joint range of motion and muscle strength. Scores range from 0 to 100, higher score indicating better function. Compare to contralateral (unaffected shoulder).
American Shoulder and Elbow Surgeon score | 6 months post op
  Evaluation criteria used to assess shoulder joint function based on the patient's pain and accumulated daily activities. Possible scores range from 0 to 100, higher scores indicating better shoulder function.
SF-12 (12-item Short Form Survey) | 6 months post op
  A general health questionnaire, drawn from the original SF-36 questionnaire. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average
University of California-Los Angeles Shoulder score | 12 months post op
  Shoulder scoring system mainly consisting of two parts. Patients subjectively evaluate pain and functional activity; and doctors objectively evaluate shoulder joint range of motion and muscle strength. Scores range from 0 to 35, with a higher score indicating a better function.
Constant-Murray Shoulder Score | 12 months post op
  Shoulder score system mainly consisting of two parts. Patients subjectively evaluate pain and activity level; doctors objectively evaluate shoulder joint range of motion and muscle strength. Scores range from 0 to 100, higher score indicating better function. Compare to contralateral (unaffected shoulder).
American Shoulder and Elbow Surgeon score | 12 months post op
  Evaluation criteria used to assess shoulder joint function based on the patient's pain and accumulated daily activities. Possible scores range from 0 to 100, higher scores indicating better shoulder function.
SF-12 (12-item Short Form Survey) | 12 months post op
  A general health questionnaire, drawn from the original SF-36 questionnaire. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average
University of California-Los Angeles Shoulder score | 24 months post op
  Shoulder scoring system mainly consisting of two parts. Patients subjectively evaluate pain and functional activity; and doctors objectively evaluate shoulder joint range of motion and muscle strength. Scores range from 0 to 35, with a higher score indicating a better function.
Constant-Murray Shoulder Score | 24 months post op
  Shoulder score system mainly consisting of two parts. Patients subjectively evaluate pain and activity level; doctors objectively evaluate shoulder joint range of motion and muscle strength. Scores range from 0 to 100, higher score indicating better function. Compare to contralateral (unaffected shoulder).
American Shoulder and Elbow Surgeon score | 24 months post op
  Evaluation criteria used to assess shoulder joint function based on the patient's pain and accumulated daily activities. Possible scores range from 0 to 100, higher scores indicating better shoulder function.
SF-12 (12-item Short Form Survey) | 24 months post op
  A general health questionnaire, drawn from the original SF-36 questionnaire. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bogard, DO, Principal Investigator — Community Memorial Health System
Locations (2):
- United States (2):
  - Community Memorial Health System, Ventura, California
  - Ventura County Medical Center, Ventura, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angeline ME, Ma R, Pascual-Garrido C, Voigt C, Deng XH, Warren RF, Rodeo SA. Effect of diet-induced vitamin D deficiency on rotator cuff healing in a rat model. Am J Sports Med. 2014 Jan;42(1):27-34. doi: 10.1177/0363546513505421. Epub 2013 Oct 16. PMID 24131579
- [Background] Oh JH, Kim SH, Kim JH, Shin YH, Yoon JP, Oh CH. The level of vitamin D in the serum correlates with fatty degeneration of the muscles of the rotator cuff. J Bone Joint Surg Br. 2009 Dec;91(12):1587-93. doi: 10.1302/0301-620X.91B12.22481. PMID 19949122
- [Background] Ryu KJ, Kim BH, Lee Y, Dan J, Kim JH. Low Serum Vitamin D Is Not Correlated With the Severity of a Rotator Cuff Tear or Retear After Arthroscopic Repair. Am J Sports Med. 2015 Jul;43(7):1743-50. doi: 10.1177/0363546515578101. Epub 2015 Apr 13. PMID 25868637
- [Background] Harada GK, Arshi A, Fretes N, Formanek B, Gamradt S, McAllister DR, Petrigliano FA. Preoperative Vitamin D Deficiency Is Associated With Higher Postoperative Complications in Arthroscopic Rotator Cuff Repair. J Am Acad Orthop Surg Glob Res Rev. 2019 Jul 3;3(7):e075. doi: 10.5435/JAAOSGlobal-D-19-00075. eCollection 2019 Jul. PMID 31579883
- [Background] Dougherty KA, Dilisio MF, Agrawal DK. Vitamin D and the immunomodulation of rotator cuff injury. J Inflamm Res. 2016 Jun 14;9:123-31. doi: 10.2147/JIR.S106206. eCollection 2016. PMID 27366101
- [Background] Maman E, Somjen D, Maman E, Katzburg S, Sharfman ZT, Stern N, Dolkart O. The response of cells derived from the supraspinatus tendon to estrogen and calciotropic hormone stimulations: in vitro study. Connect Tissue Res. 2016;57(2):124-30. doi: 10.3109/03008207.2015.1114615. Epub 2015 Dec 8. PMID 26646255
- [Background] Kearns MD, Alvarez JA, Tangpricha V. Large, single-dose, oral vitamin D supplementation in adult populations: a systematic review. Endocr Pract. 2014 Apr;20(4):341-51. doi: 10.4158/EP13265.RA. PMID 24246341
- [Background] Moon AS, Boudreau S, Mussell E, He JK, Brabston EW, Ponce BA, Momaya AM. Current concepts in vitamin D and orthopaedic surgery. Orthop Traumatol Surg Res. 2019 Apr;105(2):375-382. doi: 10.1016/j.otsr.2018.12.006. Epub 2019 Mar 8. PMID 30858042
- [Background] Entezari V, Lazarus M. Surgical Considerations in Managing Osteoporosis, Osteopenia, and Vitamin D Deficiency During Arthroscopic Rotator Cuff Repair. Orthop Clin North Am. 2019 Apr;50(2):233-243. doi: 10.1016/j.ocl.2018.10.006. PMID 30850081
- [Background] Reider B. Big D. Am J Sports Med. 2014 Jan;42(1):25-6. doi: 10.1177/0363546513516922. No abstract available. PMID 24384917